CLINICAL TRIAL: NCT01515748
Title: A Phase III, Open-labelled, Randomised Study of Neoadjuvant Docetaxel+Oxaliplatin+S-1 (DOS) + Surgery + Adjuvant S-1 Versus Surgery + Adjuvant S-1 in Patients With Resectable Advanced Gastric Cancer
Brief Title: Docetaxel+Oxaliplatin+S-1 (DOS) Regimen as Neoadjuvant Chemotherapy in Advanced Gastric Cancer
Acronym: PRODIGY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_R_05153; U1111-1127-0246 (Other: UTN); EFC13833 (Other: Sanofi)
Record Dates: First submitted 2012-01-10; First posted 2012-01-24 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; S 1 (combination); Tegafur; gimeracil; potassium oxonate; Oxonic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery + Adjuvant Chemotherapy (SC) (Other): Participants underwent surgery within 2 weeks after randomization followed by adjuvant chemotherapy with S-1 [(Gimeracil) + Oxo (Oteracil)] 40 milligrams per square meter (mg/m^2) administered orally twice daily, from Day 1 to 28 of each cycle for 1 year, and were followed-up after End-of-Treatment (EOT) until disease progression or death or study cut-off date, whichever comes first (maximum duration: up to 10 years).
  Interventions: Drug: S-1 (1-(2-tetrahydrofuryl)-5-fluorouracil + 5-chloro-2, 4-dihydroxypyridine (CDHP) (Gimeracil) + Oxo (Oteracil)
- Neoadjuvant Chemotherapy +Surgery +Adjuvant chemotherapy (CSC) (Experimental): Participants received neo-adjuvant chemotherapy with Docetaxel 50 mg/m^2 intravenously (IV) for greater than or equal to (>=)1 hour (hr) on Day 1 of each treatment cycle plus Oxaliplatin 100 mg/m^2 IV for >=2 hr on Day 1 of each treatment cycle plus S-1 [(Gimeracil) + Oxo (Oteracil)] 40 mg/m^2 administered orally twice daily from Day 1 to 14, of each treatment cycle followed by surgery approximately 1-3 weeks after completion of neo-adjuvant chemotherapy and adjuvant chemotherapy with S-1 [(Gimeracil) + Oxo (Oteracil)] 40 mg/m^2 administered orally twice daily, from Day 1 to 28 of each cycle for 1 year, and were followed-up after EOT until disease progression or death or study cut-off date, whichever comes first (maximum duration: up to 10 years).
  Interventions: Drug: Docetaxel (XRP6976); Drug: Oxaliplatin (SR96669); Drug: S-1 (1-(2-tetrahydrofuryl)-5-fluorouracil + 5-chloro-2, 4-dihydroxypyridine (CDHP) (Gimeracil) + Oxo (Oteracil)

INTERVENTIONS:
Drug: Docetaxel (XRP6976) — Pharmaceutical form:solution for infusion Route of administration: intravenous
  Arms: Neoadjuvant Chemotherapy +Surgery +Adjuvant chemotherapy (CSC)
Drug: Oxaliplatin (SR96669) — Pharmaceutical form:solution for infusion Route of administration: intravenous
  Arms: Neoadjuvant Chemotherapy +Surgery +Adjuvant chemotherapy (CSC)
Drug: S-1 (1-(2-tetrahydrofuryl)-5-fluorouracil + 5-chloro-2, 4-dihydroxypyridine (CDHP) (Gimeracil) + Oxo (Oteracil) — Pharmaceutical form:Tablet Route of administration: Oral

SUMMARY:
Primary Objective:

- To compare the 3-year progression free survival (PFS) in the two treatment arms.

Secondary Objectives:

* Overall survival (OS).
* Postoperative pathological stage and R0 (complete) resection rate.
* Safety: Toxicities associated with neoadjuvant chemotherapy, surgery, morbidity/mortality, toxicity of adjuvant chemotherapy.

DETAILED DESCRIPTION:
Participants in the neoadjuvant chemotherapy arm were treated for 3 cycles (1 cycle is 21 days) before surgery and treated for a year with S-1. Participants in the adjuvant chemotherapy arm underwent surgery and were treated for a year with S-1. All participants were followed during and after the study treatment until death or disease progression, whichever comes first.

ELIGIBILITY:
Inclusion criteria :

* Participants with new histologically confirmed, newly diagnosed, localized gastric or gastro-oesophageal adenocarcinoma, that is considered resectable.
* Participants with clinical stage (T2-3/N(+), T4/N(+/-):N positive means greater than or equal to [>=] 8 in hour axis).
* Signed informed consent.

Exclusion criteria:

* Aged less than (<) 20 years or >= 76 years. Performance status >=2 in Eastern Cooperative Oncology Group (ECOG) scale
* The participants who had the history of other malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix which had been already successfully treated.
* Previous surgery on neoplasm of stomach.
* Participants who did not completely recovered from surgery.
* Distant metastases (M1) to other organs including distant nodal groups (retropancreatic, para-aortic, portal, retroperitoneal, mesenteric node). severe/unstable angina, coronary artery bypass graft, congestive heart failure, transient ischemic attack within 6 months prior to enrollment in the study.
* Any previous palliative, adjuvant or neoadjuvant chemotherapy and/or radiotherapy and/or immunotherapy, for the currently treated gastric cancer.
* Participants with active infection or sepsis.
* Intolerance of oral taking or malabsorption: lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of S-1. Ileus, chronic inflammatory intestinal disease or extensive resection of the small intestine and other disorders which limit drug resorption. This includes gastric dumping syndrome, indications of accelerated passage through the small intestine and indications of resorption disorders after intestinal surgery.
* Greater than or equal to grade 2 severe tumour haemorrhage.
* Simultaneous participation in another study, or participation in another study within 4 weeks of commencement of this study.
* Pregnant or lactating participants.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2011-12-30 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo KANG, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Administrative Office, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kang YK, Kim HD, Yook JH, Park YK, Lee JS, Kim YW, Kim JY, Ryu MH, Rha SY, Chung IJ, Kim IH, Oh SC, Park YS, Cheong JH, Jeong O, Heo MH, Kim HK, Park C, Yoo CH, Kang SY, Zang DY, Jang YJ, Sul JY, Kim JG, Kim BS, Beom SH, Hwang JE, Ryu SW, Kook MC, Ryoo BY, Kim H, Yoo MW, Lee NS, Lee SH, Noh SH. Neoadjuvant Docetaxel, Oxaliplatin, and S-1 Plus Surgery and Adjuvant S-1 for Resectable Advanced Gastric Cancer: Updated Overall Survival Outcomes From Phase III PRODIGY. J Clin Oncol. 2024 Sep 1;42(25):2961-2965. doi: 10.1200/JCO.23.02167. Epub 2024 Jul 12. PMID 38996201
- [Derived] Kang YK, Yook JH, Park YK, Lee JS, Kim YW, Kim JY, Ryu MH, Rha SY, Chung IJ, Kim IH, Oh SC, Park YS, Son T, Jung MR, Heo MH, Kim HK, Park C, Yoo CH, Choi JH, Zang DY, Jang YJ, Sul JY, Kim JG, Kim BS, Beom SH, Cho SH, Ryu SW, Kook MC, Ryoo BY, Kim HK, Yoo MW, Lee NS, Lee SH, Kim G, Lee Y, Lee JH, Noh SH. PRODIGY: A Phase III Study of Neoadjuvant Docetaxel, Oxaliplatin, and S-1 Plus Surgery and Adjuvant S-1 Versus Surgery and Adjuvant S-1 for Resectable Advanced Gastric Cancer. J Clin Oncol. 2021 Sep 10;39(26):2903-2913. doi: 10.1200/JCO.20.02914. Epub 2021 Jun 16. PMID 34133211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 sites in Korea. A total of 693 participants were screened between 30 December 2011 to 02 January 2019, of which, 163 were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: Total of 530 participants were enrolled and randomized in study. Assignment was done using Interactive Web-Response System (IWRS) in 1:1 to treatment arms. Randomization was stratified by site and Tumor size, Lymph Nodes affected, Metastases (TNM) [T2/N+,T3-4/N+,T4/N-] stage.
Period: Overall Study
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Started (Randomized) | 264 | 266
Treated | 195 | 241
Completed | 225 | 211
Not Completed | 39 | 55
Not completed — Withdrawal by Subject | 32 | 41
Not completed — Lost to Follow-up | 2 | 4
Not completed — Other than specified above | 5 | 10

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-Treat (ITT) population which included all randomized participants.
Groups:
- Surgery + Adjuvant Chemotherapy (SC): Participants underwent surgery within 2 weeks after randomization followed by adjuvant chemotherapy with S-1 [(Gimeracil) + Oxo (Oteracil)] 40 mg/m^2 administered orally twice daily, from Day 1 to 28 of each cycle for 1 year, and were followed-up after EOT until disease progression or death or study cut-off date, whichever comes first (maximum duration: up to 10 years).
- Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC): Participants received neo-adjuvant chemotherapy with Docetaxel 50 mg/m^2 IV for >= 1 hr on Day 1 of each treatment cycle plus Oxaliplatin 100 mg/m^2 IV for >=2 hr on Day 1 of each treatment cycle plus S-1 [(Gimeracil) + Oxo (Oteracil)] 40 mg/m^2 administered orally twice daily from Day 1 to 14, of each treatment cycle followed by surgery approximately 1-3 weeks after completion of neo-adjuvant chemotherapy and adjuvant chemotherapy with S-1 [(Gimeracil) + Oxo (Oteracil)] 40 mg/m^2 administered orally twice daily, from Day 1 to 28 of each cycle for 1 year, and were followed-up after EOT until disease progression or death or study cut-off date, whichever comes first (maximum duration: up to 10 years).
- Total: Total of all reporting groups
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC) | Total
Number analyzed (Participants) | 264 | 266 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.28 (10.09) | 57.11 (10.03) | 57.19 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 59 | 109
  Male | 214 | 207 | 421
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 3-Year Progression-Free Survival (PFS), as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)1.1
Description: PFS was defined as the time from randomization to objective tumor progression, or recurrence or death. Progressive disease (PD) was defined as follows: 1) In Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC) Arm, PD was determined according to the RECIST 1.1 Criteria during the neo-adjuvant chemotherapy period; 2) Irrespective of curative resection, if an intraoperative distant metastasis was observed or a distant metastasis was reported from pathology, it was considered PD; 3) If residual cancer cells were visually identified at the resection margin during surgery but could not be completely resected (R2), it was considered PD; 4) If residual cancer cells were finally confirmed at the resection margin during postoperative histology (R1), it was considered PD; 5) In case of finding a recurrence/distant metastasis or a new lesion during follow-up after R0 complete resection, it was defined as the first tumor assessment date when it was observed.
Time Frame: 3 years
Population: Full Analysis Set (FAS): included all randomized participants who satisfied inclusion/exclusion criteria and had at least one tumor assessment after baseline visit (Day 0). The CSC Arm included all participants exposed to at least one dose of Docetaxel+Oxaliplatin+S-1 investigational products. The SC Arm included all participants who had surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 246 | 233
percentage of participants | 60.24 [53.55 to 66.28] | 66.82 [60.13 to 72.65]
Statistical Analysis 1: Comparison: Surgery + Adjuvant Chemotherapy (SC) vs Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC); Analysis was performed using Kaplan-Meier method. Comparison was stratified based on site and TNM classification (T4/N-, T2/N+, T3-4/N+); Test type: Superiority; p = 0.0152, Stratified Log Rank — Threshold for statistical significance at 0.049

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Analyzed using Kaplan-Meier method.
Time Frame: From randomization to date of death due to any cause (maximum duration: up to 10 years)
Population: Analysis was performed on FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 246 | 233
months | NA [NA to NA] — Median and upper and lower limit of confidence interval could not be calculated because of less number of participants reaching the OS event i.e., few participants died. | NA [NA to NA] — Median and upper and lower limit of confidence interval could not be calculated because of less number of participants reaching the OS event i.e., few participants died.

3. Secondary Outcome: Number of Participants With Post-Operative Pathological Stage Response
Description: TNM pathological stage was determined according to standardized histopathology and the American Joint Committee on Cancer (AJCC) staging system 7th Edition (Stages 0,IA,IB,IIA,IIB,IIIA,IIIB,IIIC and IV). Stage 0=carcinoma in situ with no metastatic potential; Stage IA=T1N0M0; Stage IB=T2N0M0,T1N1M0; Stage IIA=T3N0M0,T2N1M0,T1N2M0;Stage IIB=T4aN0M0,T3N1M0,T2N2M0,T1N3M0;Stage IIIA=T4aN1M0,T3N2M0,T2N3M0;Stage IIIB=T4bN0-1M0,T4aN2M0,T3N3M0;Stage IIIC=T4bN2-3M0, T4aN3M0 and Stage IV= distant metastases (M1) at diagnosis; where "T" denotes "tumor size" where T1: tumor invades lamina propria, muscularis mucosae, or submucosa; T2: invades muscularis propria; T3: invasion of subserosa; T4: T4a: penetrate serosa (visceral peritoneum) T4b: invade adjacent tissue and " N" denotes "nodes affected" where N1:1-2 positive lymph nodes; N2:3-6 positive lymph nodes; N3: 7 or more positive lymph nodes and "M" denotes metastases where M0: no distant metastases. Higher stages indicates worse outcome.
Time Frame: Up to 10 years
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 246 | 222
Participants
  Stage 0 | 0 | 23
  Stage IA | 9 | 32
  Stage IB | 18 | 23
  Stage IIA | 30 | 47
  Stage IIB | 25 | 36
  Stage IIIA | 35 | 18
  Stage IIIB | 49 | 24
  Stage IIIC | 46 | 14
  Stage IV | 34 | 5

4. Secondary Outcome: Percentage of Participants With R0 Resection
Description: Tumor condition was explained according to the Residual Tumor (R) Classification: R0; No residual cancer (negative cross-section), R1; Microscopically observed residual cancer (positive cross-section), R2; Macroscopically observed residual cancer.
Time Frame: Up to 10 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 246 | 222
percentage of participants | 83.74 [79.13 to 88.35] | 95.50 [92.77 to 98.22]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AE) that appeared or worsened during the treatment period (up to 30 days after the last dose of the investigational product). SAE was an AE or adverse drug reaction at any dose of the investigational product that corresponded to one of the following: resulting in death or is life threatening; requiring in-patient hospitalization or prolongation of existing hospitalization; resulting in persistent or significant disability of dysfunction; resulting in congenital anomaly or birth defect; important medical event.
Time Frame: From randomization up to 30 days after last dose of study drug (maximum duration: up to 10 years)
Population: Analysis was performed on safety population which included participants who were administered at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 195 | 241
Participants
  Any TEAE | 190 | 237
  Any treatment emergent SAE | 57 | 102
  TEAEs leading to permanent discontinuation | 11 | 25

6. Secondary Outcome: Number of Participants With Shift of Laboratory Parameters (Hematology) From Baseline Grade to Worst National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade >=3
Description: NCI-CTCAE version 4.03 was used to determine Grade(Gr),where Gr refers to severity of AE:Gr 1:mild; asymptomatic/mild symptoms; Gr 2:moderate;minimal; Gr 3:severe/medically significant; Gr 4:life-threatening consequences, Gr 5:death related to AE. Abnormal values for Hemoglobin(Hb)(Anemia) were based on Gr1:<lower limit of normal (LLN)-10.0g/dL; Gr2:<10.0-8.0g/dL; Gr3:<8.0g/dL; Gr4:life-threatening consequences;Gr5:death. Hb increased:Gr 1:increase(incr.) in >0-2g/dL above upper limit of normal(ULN);Gr2: incr. in >2-4g/dL above ULN; Gr3:incr. in >4gm/dL above ULN. White blood cell (WBC) decreased: Gr1:<LLN - 3000/mm^3;Gr2: <3000-2000/mm^3; Gr3:<2000-1000/mm^3;Gr4:<1000/mm^3. WBC (Leukocytosis):Gr3:>100,000/mm^3, Gr4:clinical manifestations of leucostasis;Gr5:Death. Abnormal Neutrophil count (ANC):- Gr1:<LLN-1500/mm^3;Gr2:<1500-1000/mm^3; Gr3: <1000-500/mm^3; Gr4:<500/mm^3. Platelet count decreased: Gr1:<LLN-75,000/mm^3;Gr2:<75,000-50,000/mm^3;Gr3:<50,000-25,000/mm^3;Gr4:<25,000/mm^3.
Time Frame: From Baseline up to 30 days after last dose of study drug (maximum duration: up to 10 years)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 195 | 241
Participants
  Hb(Anemia) Gr 0 at Baseline to Gr >=3 | 0 | 0
  Hb(Anemia) Gr 1 at Baseline to Gr >=3 | 0 | 4
  Hb(Anemia) Gr 2 at Baseline to Gr >=3 | 1 | 1
  Hb(Anemia) Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hb(Anemia) Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hb(Anemia) Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hb increased Gr 0 at Baseline to Gr >=3 | 0 | 0
  Hb increased Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hb increased Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hb increased Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hb increased Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hb increased Gr 5 at Baseline to Gr >=3 | 0 | 0
  WBC decreased Gr 0 at Baseline to Gr >=3 | 1 | 8
  WBC decreased Gr 1 at Baseline to Gr >=3 | 0 | 1
  WBC decreased Gr 2 at Baseline to Gr >=3 | 0 | 0
  WBC decreased Gr 3 at Baseline to Gr >=3 | 0 | 0
  WBC decreased Gr 4 at Baseline to Gr >=3 | 0 | 0
  WBC decreased Gr 5 at Baseline to Gr >=3 | 0 | 0
  WBC (Leukocytosis) Gr 0 at Baseline to Gr >=3 | 0 | 1
  WBC (Leukocytosis) Gr 1 at Baseline to Gr >=3 | 0 | 0
  WBC (Leukocytosis) Gr 2 at Baseline to Gr >=3 | 0 | 0
  WBC (Leukocytosis) Gr 3 at Baseline to Gr >=3 | 0 | 0
  WBC (Leukocytosis) Gr 4 at Baseline to Gr >=3 | 0 | 0
  WBC (Leukocytosis) Gr 5 at Baseline to Gr >=3 | 0 | 0
  ANC Gr 0 at Baseline to Gr >=3 | 14 | 40
  ANC Gr 1 at Baseline to Gr >=3 | 0 | 0
  ANC Gr 2 at Baseline to Gr >=3 | 1 | 0
  ANC Gr 3 at Baseline to Gr >=3 | 0 | 0
  ANC Gr 4 at Baseline to Gr >=3 | 0 | 0
  ANC Gr 5 at Baseline to Gr >=3 | 0 | 0
  Platelet count decreased Gr0 at Baseline to Gr >=3 | 0 | 5
  Platelet count decreased Gr1 at Baseline to Gr >=3 | 0 | 0
  Platelet count decreased Gr2 at Baseline to Gr >=3 | 0 | 0
  Platelet count decreased Gr3 at Baseline to Gr >=3 | 0 | 0
  Platelet count decreased Gr4 at Baseline to Gr >=3 | 0 | 0
  Platelet count decreased Gr5 at Baseline to Gr >=3 | 0 | 0

7. Secondary Outcome: Number of Participants With Shift of Laboratory Parameters (Sodium and Potassium Levels) From Baseline Grade to Worst NCI-CTCAE Grade >=3
Description: NCI-CTCAE version 4.03 was used to determine Gr,where Gr refers to severity of AE: Gr 1: mild; asymptomatic/mild symptoms; Gr 2: moderate; minimal; Gr 3:severe/medically significant; Gr 4:life-threatening consequences, Gr 5:death related to AE. Abnormal values for Sodium (Hyponatremia) were based on Gr1: <LLN-130 mmol/L; Gr3: <130-120 mmol/L; Gr4: <120 mmol/L; life-threatening consequences; Gr5: death. Sodium (Hypernatremia):Gr 1: >ULN-150 mmol/L; Gr2: >150-155 mmol/L; Gr3:>155-160 mmol/L;hospitalization; Gr4: >160 mmol/L; life-threatening consequences; Gr5: Death. Potassium (Hypokalemia): Gr 1: <LLN-3.0 mmol/L; Gr2: <LLN-3.0 mmol/L; symptomatic; intervention indicated; Gr3: <3.0-2.5 mmol/L; hospitalization indicated; Gr4: <2.5 mmol/L; life-threatening consequences; Gr5: Death; Potassium(Hyperkalemia): Gr 1: >ULN-5.5 mmol/L; Gr2: >5.5-6.0 mmol/L; Gr3: >6.0-7.0 mmol/L; hospitalization indicated; Gr4: >7.0 mmol/L; life-threatening consequences; Gr5: Death.
Time Frame: From Baseline up to 30 days after last dose of study drug (maximum duration: up to 10 years)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 195 | 241
Participants
  Hyponatremia Gr 0 at Baseline to Gr >=3 | 1 | 7
  Hyponatremia Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hyponatremia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hyponatremia Gr 3 at Baseline to Gr >=3 | 0 | 1
  Hyponatremia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hyponatremia Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hypernatremia Gr 0 at Baseline to Gr >=3 | 0 | 0
  Hypernatremia Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hypernatremia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hypernatremia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hypernatremia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hypernatremia Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hypokalemia Gr 0 at Baseline to Gr >=3 | 1 | 2
  Hypokalemia Gr 1 at Baseline to Gr >=3 | 1 | 1
  Hypokalemia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hypokalemia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hypokalemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hypokalemia Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hyperkalemia Gr 0 at Baseline to Gr >=3 | 1 | 4
  Hyperkalemia Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hyperkalemia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hyperkalemia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hyperkalemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hyperkalemia Gr 5 at Baseline to Gr >=3 | 0 | 0

8. Secondary Outcome: Number of Participants With Shift of Laboratory Parameters (Calcium, Creatinine and Albumin Levels) From Baseline Grade to Worst NCI-CTCAE Grade >=3
Description: NCI-CTCAE version 4.03 was used to determine Gr,where Gr refers to severity of AE:Gr 1:mild; asymptomatic/mild symptoms; Gr 2:moderate;minimal; Gr 3:severe/medically significant; Gr 4:life-threatening consequences, Gr 5:death related to AE. Abnormal values for Calcium(Hypocalcemia) were based on Gr1: Corrected serum calcium of <LLN-8.0 mg/dL; Gr2: Corrected serum calcium of <8.0-7.0 mg/dL; Gr3: Corrected serum calcium of <7.0-6.0 mg/dL ; Gr4: Corrected serum calcium of <6.0 mg/dL;Gr5:death. Calcium(Hypercalcemia):Gr 1: Corrected serum calcium of >ULN -11.5 mg/dL; Gr2: Corrected serum calcium of >11.5-12.5 mg/dL; Gr3: Corrected serum calcium of >12.5-13.5 mg/dL; Gr4: Corrected serum calcium of >13.5 mg/dL;Gr5:Death. Creatinine increased: Gr 1: >1-1.5*baseline; >ULN-1.5*ULN; Gr2: >1.5-3.0*baseline; >1.5-3.0*ULN; Gr3: >3.0 baseline; >3.0-6.0*ULN; Gr4: >6.0 x ULN. Albumin(Hypoalbuminemia): Gr 1: <LLN-3 g/dL; Gr2: <3-2 g/dL; Gr3: <2 g/dL; Gr4:life-threatening consequences;Gr5:Death.
Time Frame: From Baseline up to 30 days after last dose of study drug (maximum duration: up to 10 years)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 195 | 241
Participants
  Hypocalcemia Gr 0 at Baseline to Gr >=3 | 1 | 0
  Hypocalcemia Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hypocalcemia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hypocalcemia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hypocalcemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hypocalcemia Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hypercalcemia Gr 0 at Baseline to Gr >=3 | 1 | 1
  Hypercalcemia Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hypercalcemia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hypercalcemia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hypercalcemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hypercalcemia Gr 5 at Baseline to Gr >=3 | 0 | 0
  Creatinine increased Gr 0 at Baseline to Gr >=3 | 4 | 8
  Creatinine increased Gr 1 at Baseline to Gr >=3 | 0 | 0
  Creatinine increased Gr 2 at Baseline to Gr >=3 | 0 | 0
  Creatinine increased Gr 3 at Baseline to Gr >=3 | 0 | 0
  Creatinine increased Gr 4 at Baseline to Gr >=3 | 0 | 0
  Creatinine increased Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hypoalbuminemia Gr 0 at Baseline to Gr >=3 | 1 | 2
  Hypoalbuminemia Gr 1 at Baseline to Gr >=3 | 0 | 0
  Hypoalbuminemia Gr 2 at Baseline to Gr >=3 | 0 | 0
  Hypoalbuminemia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hypoalbuminemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hypoalbuminemia Gr 5 at Baseline to Gr >=3 | 0 | 0

9. Secondary Outcome: Number of Participants With Shift of Laboratory Parameters (Aspartate Aminotransferase, Alanine Aminotransferase,Blood Bilirubin,Alkaline Phosphatase and Glucose Levels) From Baseline Grade to Worst NCI-CTCAE Grade >=3
Description: NCI-CTCAE version 4.03 was used to determine Gr, where Gr refers to severity of AE: Gr 1:mild; asymptomatic/mild symptoms; Gr 2:moderate; minimal; Gr 3:severe/medically significant; Gr 4:life-threatening consequences, Gr 5:death related to AE. Abnormal values for Aspartate and alanine aminotransferase increased were based on Gr1: >ULN-3.0*ULN; Gr2: >3.0-5.0*ULN; Gr3: >5.0-20.0*ULN; Gr4: >20.0*ULN. Blood bilirubin increased: Gr1: >ULN-1.5*ULN; Gr2 >1.5-3.0*ULN; Gr3: >3.0-10.0*ULN; Gr4: >10.0*ULN. Alkaline phosphatase increased: Gr1: >ULN-2.5*ULN; Gr2: >2.5-5.0*ULN; Gr3: >5.0-20.0*ULN; Gr4: >20.0*ULN. Glucose (Hypoglycemia): Gr 1: <LLN-55 mg/dL; Gr2: <55-40 mg/dL;Gr3: <40-30 mg/dL; Gr4: <30 mg/dL; Gr5:Death. Glucose (Hyperglycemia): Gr 1: Fasting glucose value >ULN-160 mg/dL; Gr2: Fasting glucose value >160-250 mg/dL; Gr3: >250-500 mg/dL; Gr4: >500 mg/dL; Gr5: Death.
Time Frame: From Baseline up to 30 days after last dose of study drug (maximum duration: up to 10 years)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 195 | 241
Participants
  Aspartate aminotransferase Gr0 at Baseline toGr>=3 | 1 | 1
  Aspartate aminotransferase Gr1 at Baseline toGr>=3 | 0 | 0
  Aspartate aminotransferase Gr2 at Baseline toGr>=3 | 0 | 0
  Aspartate aminotransferase Gr3 at Baseline toGr>=3 | 0 | 0
  Aspartate aminotransferase Gr4 at Baseline toGr>=3 | 0 | 0
  Aspartate aminotransferase Gr5 at Baseline toGr>=3 | 0 | 0
  Alanine aminotransferase Gr0 at Baseline to Gr >=3 | 0 | 1
  Alanine aminotransferase Gr1 at Baseline to Gr >=3 | 0 | 0
  Alanine aminotransferase Gr2 at Baseline to Gr >=3 | 0 | 0
  Alanine aminotransferase Gr3 at Baseline to Gr >=3 | 0 | 0
  Alanine aminotransferase Gr4 at Baseline to Gr >=3 | 0 | 0
  Alanine aminotransferase Gr5 at Baseline to Gr >=3 | 0 | 0
  Bilirubin increased Gr 0 at Baseline to Gr >=3 | 2 | 4
  Bilirubin increased Gr 1 at Baseline to Gr >=3 | 1 | 0
  Bilirubin increased Gr 2 at Baseline to Gr >=3 | 1 | 0
  Bilirubin increased Gr 3 at Baseline to Gr >=3 | 0 | 0
  Bilirubin increased Gr 4 at Baseline to Gr >=3 | 0 | 0
  Bilirubin increased Gr 5 at Baseline to Gr >=3 | 0 | 0
  Alkaline phosphatase Gr 0 at Baseline to Gr >=3 | 3 | 0
  Alkaline phosphatase Gr 1 at Baseline to Gr >=3 | 0 | 0
  Alkaline phosphatase Gr 2 at Baseline to Gr >=3 | 0 | 0
  Alkaline phosphatase Gr 3 at Baseline to Gr >=3 | 0 | 0
  Alkaline phosphatase Gr 4 at Baseline to Gr >=3 | 0 | 0
  Alkaline phosphatase Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hypoglycemia Gr 0 at Baseline to Gr >=3 | 4 | 0
  Hypoglycemia Gr 1 at Baseline to Gr >=3 | 1 | 0
  Hypoglycemia Gr 2 at Baseline to Gr >=3 | 1 | 0
  Hypoglycemia Gr 3 at Baseline to Gr >=3 | 0 | 0
  Hypoglycemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hypoglycemia Gr 5 at Baseline to Gr >=3 | 0 | 0
  Hyperglycemia Gr 0 at Baseline to Gr >=3 | 4 | 12
  Hyperglycemia Gr 1 at Baseline to Gr >=3 | 13 | 13
  Hyperglycemia Gr 2 at Baseline to Gr >=3 | 2 | 10
  Hyperglycemia Gr 3 at Baseline to Gr >=3 | 3 | 2
  Hyperglycemia Gr 4 at Baseline to Gr >=3 | 0 | 0
  Hyperglycemia Gr 5 at Baseline to Gr >=3 | 0 | 0

10. Secondary Outcome: Number of Participants With Shift of Laboratory Parameters (Creatinine Clearance [Chronic Kidney Disease]) From Baseline Grade to Worst NCI-CTCAE Grade >=3
Description: NCI-CTCAE version 4.03 was used to determine Gr, where Gr refers to severity of AE: Gr 1: mild; asymptomatic/mild symptoms; Gr 2: moderate; minimal; Gr 3: severe/medically significant; Gr 4:life-threatening consequences, Gr 5:death related to AE. Abnormal values for Creatinine Clearance(Chronic kidney disease) were based on: Gr 1: estimated glomerular filtration rate (eGFR) or creatinine clearance (CrCl) <LLN-60ml/min/1.73 m^2; Gr2: eGFR or CrCl 59-30 ml/min/1.73 m^2; Gr3: eGFR or CrCl 29-15 ml/min/1.73 m^2; Gr4: eGFR or CrCl <15 ml/min/1.73 m^2; Gr5: Death.
Time Frame: From Baseline up to 30 days after last dose of study drug (maximum duration: up to 10 years)
Population: Analysis was performed on safety population. Data was planned to be collected and analyzed for Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC) arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
Number analyzed (Participants) | 241
Participants
  Creatinine Clearance Gr 0 at Baseline to Gr >=3 | 0
  Creatinine Clearance Gr 1 at Baseline to Gr >=3 | 0
  Creatinine Clearance Gr 2 at Baseline to Gr >=3 | 0
  Creatinine Clearance Gr 3 at Baseline to Gr >=3 | 0
  Creatinine Clearance Gr 4 at Baseline to Gr >=3 | 0
  Creatinine Clearance Gr 5 at Baseline to Gr >=3 | 0

ADVERSE EVENTS:
Time Frame: AE data was collected from the time of signed informed consent to 30 days following the last administration of study treatment (maximum duration: up to 10 years)
Description: All-Cause Mortality data collected during the study was assessed for all randomized population. SAE and other AE data was assessed for safety population. Disease progression related death were not reported as AE.
Arm/Group | Surgery + Adjuvant Chemotherapy (SC) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC)
All-Cause Mortality (participants affected / at risk) | 91/264 | 78/266
Serious Adverse Events (participants affected / at risk) | 57/195 | 102/241
Other Adverse Events (participants affected / at risk) | 141/195 | 201/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery + Adjuvant Chemotherapy (SC) (N=195) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC) (N=241)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 21 (23)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic Infarction (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 12 (13)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 6 (7) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6) | 4 (4)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-Abdominal Fluid Collection (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ischaemic Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical Ileus (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (1) | 3 (5)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 4 (4)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal Infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Large Intestine Infection (Infections and infestations) | 0 (0) | 1 (1)
Lung Abscess (Infections and infestations) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Afferent Loop Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic Leak (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Gastrointestinal Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripancreatic Fluid Collection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 1 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Finger Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery + Adjuvant Chemotherapy (SC) (N=195) | Neoadjuvant Chemotherapy +Surgery +Adjuvant Chemotherapy (CSC) (N=241)
Anaemia (Blood and lymphatic system disorders) | 19 (20) | 18 (21)
Dry Eye (Eye disorders) | 11 (11) | 8 (10)
Lacrimation Increased (Eye disorders) | 23 (27) | 22 (25)
Abdominal Pain Upper (Gastrointestinal disorders) | 7 (7) | 14 (16)
Dyspepsia (Gastrointestinal disorders) | 43 (65) | 65 (90)
Influenza Like Illness (General disorders) | 16 (19) | 18 (21)
Nasopharyngitis (Infections and infestations) | 12 (13) | 21 (24)
Alanine Aminotransferase Increased (Investigations) | 20 (23) | 18 (20)
Aspartate Aminotransferase Increased (Investigations) | 21 (24) | 20 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 33 (42)
Headache (Nervous system disorders) | 4 (5) | 20 (28)
Neuropathy Peripheral (Nervous system disorders) | 2 (3) | 18 (20)
Peripheral Sensory Neuropathy (Nervous system disorders) | 8 (9) | 42 (55)
Insomnia (Psychiatric disorders) | 12 (12) | 30 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 21 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 14 (17)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 20 (25)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 117 (122)
Nail Ridging (Skin and subcutaneous tissue disorders) | 6 (6) | 19 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (31) | 37 (53)
Rash (Skin and subcutaneous tissue disorders) | 10 (13) | 11 (12)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 52 (54) | 49 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT01515748/Prot_002.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT01515748/SAP_003.pdf